CLINICAL TRIAL: NCT01753843
Title: A Randomised Controlled Trial to Evaluate the Role of Brief Delay in Cord Clamping in Preterm Neonates (34-36weeks) on Short Term Neurodevelopmental Outcome
Brief Title: Brief Delay in Cord Clamping and Neurobehaviour in Preterms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, Principal Investigator, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Brief Delay in Cord Clamping
Record Dates: First submitted 2012-12-18; First posted 2012-12-20 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Preterm Birth
Keywords: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early cord clamping (Active Comparator): cord clamping within 20 sec
  Interventions: Procedure: early cord clamping
- brief delay in cord clamping (Experimental): cord clamping delayed by 30 to 60 seconds
  Interventions: Procedure: Brief Delay in cord clamping

INTERVENTIONS:
Procedure: early cord clamping — early ( <20 seconds)
  Arms: early cord clamping
Procedure: Brief Delay in cord clamping — delay in cord clamping 30 to 60 seconds
  Arms: brief delay in cord clamping

SUMMARY:
RESEARCH HYPOTHESIS Brief delay(>30 sec to <60 sec ) in cord clamping as compared to early cord clamping (< 20 sec) leads to a better short term neurobehavioural outcome in preterm (34-36 wks) neonates when assessed by neurobehavioral assessment of preterm infants (n.a.p.i.) at 37 weeks of post conceptional age

DETAILED DESCRIPTION:
Delayed cord clamping (DCC) : Well described phenomenon in term infants .

* The optimal timing of clamping of umbilical cord in preterm infants : A subject of debate.
* Even a brief delay in cord clamping leads to an additional transfer of iron amounting to 40-50 mg/kg which may prevent iron deficiency.¹
* This low cost intervention can have significant public health importance in resource constrained settings.
* The effect of this intervention on neurobehaviour of preterm neonates has not been assessed.
* This aspect has been identified by WHO and Cochrane as a potentially researchable area

ELIGIBILITY:
Inclusion Criteria:

* All preterm deliveries -infants born at 34 weeks 0 days to 36 weeks +6 days gestational age as estimated by last menstrual period or early ultrasound scan.
* Infants delivered vaginally or by caesarean section in cephalic presentation
* Singleton pregnancy
* Parental consent

Exclusion Criteria:

* Fetus with gross congenital anomaly
* Fetus with hydrops
* Rh negative pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
short term neurobehavioral outcome | at 37 weeks post conceptional age
  using N.A.P.I (neurobehavioural assessment of preterm infant)

SECONDARY OUTCOMES:
measuring cord hematocrit | at birth

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Datta, M.D., Principal Investigator — Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India